CLINICAL TRIAL: NCT02776423
Title: Transurethral Polyacrylamide Hydrogel Injection in Patients Ineligible for Midurethral Sling Surgery
Brief Title: Polyacrylamide Injection in Patients Ineligible for Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Daniel Altman, Associate professor, Karolinska Institutet
Other Study IDs: SUGM
Record Dates: First submitted 2016-05-14; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Bulkamid; polyacrylamide gels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bulkamid — The procedure was standardized, identical for all patients, and entirely performed in an outpatient setting. All injections were performed by a single urogynecologist. Before injection all patients received a single dose trimethoprim (Idotrim®, Orion Pharma). The patient was placed in a supine position and given intraurethral topical 2% lidocaine hydrochloride gel (Xylocain®, Astra Zeneca) for anesthetic. Using a video-urethroscope and a 23-gauge needle, polyacrylamide hydrogel deposits of 0.3-0.4 mL were injected at 12, 4 and 8 o´clock into the submucosa approximately 1 cm from the bladder neck. Patients were discharged after successful voiding.
  Other Names: Polyacrylamide hydrogel

SUMMARY:
Transurethral injection using polyacrylamide hydrogel (Bulkamid®, Contura A/S, Denmark) is an established treatment for stress urinary incontinence. The rates of women reporting improvement or cure after Bulkamid injection for stress urinary incontinence range between 64-77% with a very low morbidity. However, the indications for use are unclear. Although transurethral polyacrylamide hydrogel injection is inferior to midurethral slings with regard to expected cure rates, the procedure is associated with very low rates of adverse events in general and serious adverse event in particular. As such, it may be an important alternative for patients where surgery is not considered a safe option either because of co-morbidity or because of complicated incontinence. The investigators performed a prospective study to determine the effects of transurethral polyacrylamide hydrogel injection in patients considered ineligible for midurethral sling surgery.

DETAILED DESCRIPTION:
In this prospective observational study the investigators included female patients who received treatment with transurethral polyacrylamide hydrogel injection (Bulkamid®). Patients were considered ineligible for surgery based on significant co-morbidity, one or more previously failed invasive treatments, complex urinary incontinence, or previous pelvic radiation therapy. At the baseline visit patients underwent a routine gynecological exam including pelvic ultrasonography. Patients completed validated questionnaires at the baseline visit and follow-up for evaluation of subjective treatment success. At baseline, women were asked to self-report any concomitant diseases or health conditions which were noted in the patient records together with a standard gynecological, urological and general health history. Follow-up visits were scheduled at 2 and 6 months after first injection at which time a second injection was administered at patients' discretion.

ELIGIBILITY:
Inclusion Criteria:

* Women with stress urinary incontinence considered ineligible for surgery based on significant co-morbidity, one or more previously failed invasive treatments, complex urinary incontinence, or previous pelvic radiation therapy.

Exclusion Criteria:

* Patients who do not want treatment or to participate in study follow-up
* Below 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study we included 81 female patients who received treatment with transurethral polyacrylamide hydrogel injection (Bulkamid®). Patients were considered ineligible for surgery based on significant co-morbidity, one or more previously failed invasive treatments, complex urinary incontinence, or previous pelvic radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Urinary distress inventory (UDI) overall score | 6 months

SECONDARY OUTCOMES:
UDI stress score | 6 months
UDI irritative score | 6 months
UDI obstructive score | 6 months
Adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Altman, MD, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altman D, Ghilotti F, Bellocco R, Zetterstrom J, Kopp Kallner H. Transurethral Polyacrylamide Hydrogel Injection Therapy in Women Not Eligible for Midurethral Sling Surgery. Female Pelvic Med Reconstr Surg. 2017 Sep/Oct;23(5):318-323. doi: 10.1097/SPV.0000000000000385. PMID 28106655